CLINICAL TRIAL: NCT05854329
Title: The Effects of Preoperative Immersive and Non-Immersive Virtual Reality Exposure on Dental Anxiety in Children: a Randomised Controlled Trial
Brief Title: The Effects of Preoperative Immersive and Non-Immersive Virtual Reality Exposure on Dental Anxiety in Children:A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DF CD2313/0024 (P)
Record Dates: First submitted 2023-04-21; First posted 2023-05-11 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: Immersive and Non immersive Virtual Reality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immersive Virtual Reality Exposure (Experimental): Immersive Virtual Reality Dental Game for 15 minutes. Participants will be actively involved with the game, in placing restorations, scaling virtually playing the role of the dentist.
  Interventions: Behavioral: Virtual Reality Exposure
- Non-Immersive Virtual Reality Exposure (Active Comparator): Participants will be made to watch dental related cartoon passively while sitting using the Virtual Reality device for 15 minutes.
  Interventions: Behavioral: Virtual Reality Exposure
- Control Group (No Intervention): Participants will be waiting for 15 minutes as usual prior to their treatment.

INTERVENTIONS:
Behavioral: Virtual Reality Exposure — Virtual Reality device using the immersive dental game.
  Arms: Immersive Virtual Reality Exposure; Non-Immersive Virtual Reality Exposure

SUMMARY:
The goal of this randomised controlled trial is to compare the effects of Immersive Virtual Reality(IVRE) and Non-Immersive Virtual Reality(NIVRE) andin children having dental anxiety.The main question[s] it aims to answer are:

1. Is there a significant difference in baseline dental anxiety scores, as measured using the Malay-MCDASf and PR across the IVRE, NIVRE, and control groups?
2. What is the mean change score in dental anxiety measured using the Malay-MCDASf and PR for IVRE, NIVRE, and control groups after the operative procedure?
3. Is there a significant difference in mean change score of dental anxiety measured using the Malay-MCDASf and PR across the IVRE, NIVRE, and control groups?
4. Is there a significant correlation between the Malay-MCDASf scores (subjective) and PR scores (objective) at preoperative, postoperative, and using the score changes for all groups?

DETAILED DESCRIPTION:
Participants will be randomised into three groups, Immersive Virtual Reality, Non Immersive Virtual Reality and Control Group.Immersive Virtual Reality group will be asked to play with an immersive virtual reality dental game using Virtual reality device preoperatively after which they will undergo treatment. For the Non Immersive Virtual Reality participants will be asked to watch a dental cartoon using the virtual reality device passively before treatment and the control group of no intervention, to wait as usual before treatment. All groups will undergo dental treatment of resin based fissure sealant placement under cotton roll isolation in one permanent molar.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-12 years old.
* Children who can understand and complete the Malay-MCDASf questionnaire with a score of 19 and above.
* Children who requires fissure sealants on sound permanent tooth.

Exclusion Criteria:

* Children requiring emergency dental treatment for pain, trauma or facial cellulitis.
* Children that have undergone invasive dental treatment such as extraction and pulp therapy in the past 6 months.
* Children with hearing or visual impairment, developmental or intellectual disability, cognitive impairment, balance disorders such as vertigo and cybersickness, sensitivity to the motion or flash light, having accident in the eye, face, neck or arms, history of epileptic seizures, history of cardiac problems
* Parents who refuse to allow their children to participate in the trial.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Malay-MCDASf score | 10 minutes prior to Intervention and immediately after intervention followed by dental treatment on the same day
  Malay translated Modified Child Dental Anxiety Scale faces version

SECONDARY OUTCOMES:
Change in Pulse Rate | 10 minutes prior to Intervention and immediately after intervention followed by dental treatment on the same day
  Will be measured using Pulse Oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Leezallini Selvaraj, Principal Investigator — Faculty of Dentistry Medical Ethics Committee (FDMEC)
Locations (1):
- Faculty of Dentistry, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selvaraj L, Yusof ZYM, Zakaria NN, Azizi NZ, Aalam NZ. Effects of Preoperative Immersive and Non-Immersive Virtual Reality Exposure on Dental Anxiety in Children: A Randomised Controlled Trial. Int J Paediatr Dent. 2025 Dec 22. doi: 10.1111/ipd.70066. Online ahead of print. PMID 41429659